CLINICAL TRIAL: NCT06700109
Title: INJECTABLE COLD ENERGY THERAPY FOR THE MANAGEMENT OF CHRONIC PAIN ASSOCIATED WITH OSTEOARTHRITIS OF THE KNEE: A MULTI-CENTER, RANDOMIZED, CONTROLLED STUDY (ICE STUDY)
Brief Title: INJECTABLE COLD ENERGY THERAPY FOR THE MANAGEMENT OF CHRONIC PAIN ASSOCIATED WITH OSTEOARTHRITIS OF THE KNEE
Acronym: ICE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brixton Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BXT-786-KPM-03
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: osteoarthritis; knee pain; osteoarthritis of the knee; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: MULTI-CENTER, RANDOMIZED, CONTROLLED STUDY
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Neural Ice injections (Experimental): This therapy will be injected around the superolateral, superomedial, and inferomedial genicular nerves.
  Interventions: Device: Neural Ice
- Corticosteroid injection (Active Comparator): Intraarticular corticosteroid injection is defined as a single dose of Triamcinolone 40mg injected directly into the joint space.
  Interventions: Drug: Triamcinolone acetate

INTERVENTIONS:
Device: Neural Ice — This therapy will be injected around the superolateral, superomedial, and inferomedial genicular nerves.
  Arms: Neural Ice injections
Drug: Triamcinolone acetate — A single dose of Triamcinolone 40mg injected directly into the joint space.
  Arms: Corticosteroid injection

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of Neural Ice for pain management associated with knee osteoarthritis in adults aged 22-80 years. Participants will attend study visits and complete subject diaries. Participants will be followed for 6 months after study procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 to 80, inclusive of any gender
2. Baseline pain intensity of >/= 5 of the Numeric Rating Scale (NRS) despite current treatment Confidential Brixton Biosciences Inc. Page 12 of 53 Version: 1.1, 30 August 2024
3. Chronic symptomatic osteoarthritis of the knee (K-L stage 2, 3, or 4) on plain x-rays obtained within the previous 12 months
4. At least 3 months of previous conservative treatments (NSAID, acetaminophen, physical therapy, cortisone injections) that are not currently providing relief
5. Agree to see one doctor (study investigator) for knee pain during the study period
6. Willing/able to understand the informed consent form and provide written informed consent
7. Able to complete outcome measures (including electronic patient reported outcome measures)

Exclusion Criteria:

1. Known allergy to glycerol, hyaluronic acid, poloxamer 407, or phosphate buffered saline
2. History of cryoglobulinemia
3. History of cold-induced auto-immune hemolytic anemia (e.g. paroxysmal cold hemoglobinuria or cold agglutinin disease)
4. History of cold urticaria
5. History of Chilblain's (pernio) disease in the lower extremities
6. History of Raynaud's disease
7. Open and/or infected wounds or active tumor at or near the treatment site
8. History of vascular surgery involving femoral vessels on the injection side
9. History of surgical procedures to affected limb that, in the opinion of the investigator, could have impacted the integrity of the genicular nerves or blood vessels
10. Active bacterial or fungal infection that at the discretion of the investigator would preclude study participation
11. Currently taking >60 MME/day, as determined per MDcalc.com (opioid conversion calculator)
12. History of History of systemic inflammatory conditions such as rheumatoid arthritis
13. Bleeding disorders anticoagulant therapy, unless appropriately stopped or reversed for the procedure
14. Any condition or circumstance that would impact or confound assessment of safety and/or pain. For example, comorbid or concomitant pain conditions, pre-existing lower limb neurologic deficits, any psychiatric or neurologic disease
15. Cryoneurolysis, thermal or pulsed radiofrequency ablation, or phenol injection for the index knee within the past 12 months
16. Use of intra-articular injection of corticosteroid within the previous 3 months, or hyaluronic acid, prolotherapy, Confidential Brixton Biosciences Inc. Page 13 of 53 Version: 1.1, 30 August 2024 autologous blood, or platelet rich plasma injections for the index knee within the previous 6 months
17. Known contraindication to use of a regional anesthetic block
18. Pregnant, nursing or intent of becoming pregnant during the study period
19. Any condition (such as history of significant cardiovascular, renal failure/dialysis, hepatic or other systemic comorbidity/chronic pain condition) or circumstance that, in the opinion of the investigator, would compromise the safety of the subject or the quality of study data
20. Body habitus/knee anatomy that would preclude the use of the product injection needle size
21. Participation in any clinical study of a therapeutic investigational product within 30 days prior to enrollment
22. Unwilling to refrain from participation in any other clinical study through the duration of this study
23. Unwilling to refrain from any scheduled surgeries during the duration of this study

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness | 3 months
  The proportion of subjects whose knee pain following activity (Timed Up and Go test) is reduced by ≥30% based on the NRS scale at 3 months post treatment.
Primary Safety | 6 months
  Aggregate serious device-related adverse events through final follow up visit.

SECONDARY OUTCOMES:
Secondary Effectiveness | 6 months
  The proportion of subjects whose knee pain following activity (Timed Up and Go test) is reduced by ≥30% based on the NRS scale at 6 months post treatment.
NRS Scores | 6 months
Pain medication usage | 6 months
PGIC scores | 6 months
KOOS, JR scores | 6 months
Onset of pain relief defined as pain reduced by 30% based on NRS score from baseline | 6 months
Change in Timed-Up and Go (TUG) test scores from baseline | 6 months

OTHER OUTCOMES:
Patient-Specific Functional Scale (PSFS) | 6 months
Knee procedures specific Healthcare Utilization Data | 6 months
EQ-5D-5L Global Quality of Life measure | 6 months

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Marin Health, Larkspur, California
  - Centers for Advanced Orthopedics, Washington D.C., District of Columbia
  - The Orthopaedic Institute, Gainesville, Florida
  - Emory University, Johns Creek, Georgia
  - Insight Hospital and Medical Center Chicago, Chicago, Illinois
  - NextStage Clinical Research Advanced Orthopaedic Associates, Wichita, Kansas
  - Ochsner Health System, New Orleans, Louisiana
  - NextStage Clinical Research Regenerative Orthopedics and Sports Medicine, North Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Insight Research Institute, Flint, Michigan
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - NextStage Clinical Research The Orthopedic Center, Tulsa, Oklahoma
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - NextStage Clinical Research All-American Orthopedic & Sports Medicine Institute, Houston, Texas
  - UT San Antonio, San Antonio, Texas